CLINICAL TRIAL: NCT02035410
Title: Phase 1 Study of Prevention of Cardiac Device Implantation Site Infection
Brief Title: Decrease Implantation Site INFECTION (DISINFECTION I): a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, ph.D, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DISINFECTION I
Record Dates: First submitted 2014-01-12; First posted 2014-01-14 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Infection
Keywords: cardiac devices; prevention; infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrogen peroxide pretreatment group (Active Comparator): Hydrogen peroxide pretreatment perform before cardiac devices Implantation. It disinfects the cardiac devices pocket using Hydrogen peroxide gauze.
  Interventions: Procedure: Hydrogen peroxide pretreatment group
- Control group (No Intervention): No intervention group

INTERVENTIONS:
Procedure: Hydrogen peroxide pretreatment group — Hydrogen peroxide pretreatment perform before cardiac devices Implantation. It disinfects the cardiac devices pocket using Hydrogen peroxide gauze.
  Arms: Hydrogen peroxide pretreatment group

SUMMARY:
Cardiovascular implantable electronic device (CIED) infections have been increasing out of proportion to the number of devices implanted We investigated recent trends and possible causes of the increasing numbers of Cardiovascular implantable electronic device infections.

DETAILED DESCRIPTION:
There are many studies on the preventive use of Antibiotics or povidone iodine to Cardiovascular implantable electronic device (CIED) infections.

But, studies of prophylactic use of hydrogen peroxide is still limited.

We had planned research on effects of preventive using hydrogen peroxide before cardiac devices insertion.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cardiac devices Implantation

Exclusion Criteria:

* under the age of 18
* Hydrogen peroxide allergy
* take an antibiotic
* History of infection within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2013-12; Primary Completion 2019-08 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
freedom of cardiac device-related infection | 1 year after precedure
  check the symptoms of infection. If have symptoms of infection : check the fever, heart rate, respiration rate, blood test, EKG

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seog Oh, Ph.D, Study Chair — Seoul St. Mary's Hospital
Locations (1):
- Seoul St Mary's Hospital, Seoul, Seo Ch-gu, South Korea

IPD SHARING:
Plan to Share IPD: No